CLINICAL TRIAL: NCT02416752
Title: Effect of Remifentanil on the Recovery Profile After Prolonged Head and Neck Surgery
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Suhitharan Thangavelautham, Senior resident, Singapore General Hospital
Other Study IDs: Remi 2011/421/D SGH
Record Dates: First submitted 2015-04-07; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Pain; Head and Neck Disorder
Keywords: remifentanil; head and neck surgery; recovery pofile; Opioid induced hyperalgesia; post operative pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Remifentanil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- remifentanil group: Group received intra op remifentanil infusion
  Interventions: Drug: Remifentanil
- conventional opioid gropup: Group received only conventional opioids and No infusion of remifentanil
  Interventions: Drug: choice of intra-operative opioids were left to the discretion of anesthesiologist

INTERVENTIONS:
Drug: Remifentanil — The remifentanil infusion was used intra operatively in remifentanil group and intermittent boluses of morphine or fentanyl administered for conventional opioid group
  Groups: remifentanil group
Drug: choice of intra-operative opioids were left to the discretion of anesthesiologist
  Groups: conventional opioid gropup

SUMMARY:
Opioid tolerance in the perioperative period is inevitable especially with ultra-short acting agents such as remifentanil. Existing evidence had shown that opioid induced hyperalgesia due to neuroplastic changes in the central as well as peripheral nervous system leads to sensitization of pro-nociceptive pathways. However there has been a controversy of occurrence of such tolerance following the use of remifentanil and the quality of recovery as compared to conventional opioids. The investigators evaluated the occurrence of opioid tolerance and other significant adverse effects with remifentanil in subjects undergoing head and neck surgeries. The investigators studied ASA physical status I and II adult subjects undergoing elective head and neck procedures, under general anesthesia with minimum expected duration of 2 hours. The remifentanil infusion was used in one group and intermittent boluses of morphine or fentanyl administered in another group. They were evaluated for immediate post-operative pain by using numerical rating scale (NRS), the opioid consumption, post-operative nausea, vomiting, other significant adverse effects of remifentanil and the time to discharge from PACU.

DETAILED DESCRIPTION:
We have studied 222 of you between the age of 21 and 80 years, over a period of 2 years at Singapore General Hospital, Singapore. All of you were ASA I to II and scheduled for elective head and neck surgery with minimum expected duration of 2 hours, requiring general anesthesia. The methodology of this observational study was approved by the International review Board at Singapore General Hospital, Singapore. Informed consent was obtained from you prior to the procedure. If you had previous history of either drug or alcohol abuse, have been using opioids for long term, mental disorder with difficult to understand pain scoring system, ASA physical status of III and above, your surgical procedure warranting elective postoperative ventilation you would have been excluded from this study. The study was not randomized and the choice of intra-operative opioids were left to the discretion of anesthesiologist attending you.

You were not premedicated and instructed about 11 point numerical rating score after reaching induction room. Upon arrival in the operating room, you were monitored with EKG, non-invasive arterial pressure and pulse oxymetry. The attending anesthesiologist gave you either Remifentanil or conventional opioids at standard doses from the induction of anesthesia to end of surgery. Sevoflurane, desflurane or isoflurane with oxygen air mixture were utilized to maintain anesthesia at the minimum alveolar concentration of 0.8 to 1.2 . Choice of opioid, volatile agent, muscle relaxants, airway was left to the discretion of the anesthesiologist attending the patient. Parameters including type of volatile anesthetic agent, method of air way establishment, the duration of surgery, the remifentanil used (microgram.kg-1 ) and amount of morphine or fentanyl (microgram.kg-1) were documented. Upon arrival to the PACU you were assessed for the pain.

For the first 15 minutes behavioral score (0 - calm patient with no verbal or behavioral manifestation of pain, 1 - behavioral or verbal expression of pain, and 2 - intense behavioral or verbal manifestation [crying or extreme agitation]) were utilized and subsequently numerical rating scale (NRS) was used for every 5 minutes until discharge from the PACU.

Intravenous morphine or fentanyl was used to treat immediate post-operative pain in PACU till the NRS is less than or equal to 3 as per PACU acute pain management protocol. Maximum NRS of pain, amount of morphine or fentanyl used for rescue analgesia, occurrence of either nausea or vomiting and the antiemetic used was gathered every 15 minutes. Upon discharge from the PACU, total opioids consumed, duration of the PACU (defined by time since admission to decision made for discharge by PACU anesthesiologists, to rule out the prolong PACU stay from other reasons) and occurrence of other potential side effects that affect the quality of recovery such as drowsy, nausea, vomiting, shivering and evidence of respiratory suppression ( desaturation or bradypnea ) were documented.

Our primary outcome was amount of opioids used in PACU and the secondary outcomes were the duration of PACU stay and the adverse effects of remifentanil that influence the recovery as stated above.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASA I to II, scheduled for elective head and neck surgery with minimum expected duration of 2 hours, requiring general anesthesia

Exclusion Criteria:

previous history of either drug or alcohol abuse those who have been using opioids for long term mental disorder with difficult to understand pain scoring system ASA physical status of III and above surgical procedure warranting elective postoperative ventilation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We studied 222 adult subjects between 21 and 80 years, over two years at Singapore General Hospital, Singapore. All subjects were ASA I to II and scheduled for elective head and neck surgery with minimum expected duration of 2 hours, requiring general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Amount of opioids used in PACU in morphine equivalent | 90 minutes
  average time spent in PACU

SECONDARY OUTCOMES:
Duration of PACU | 90 minutes
  average time spent in PACU
Adverse effects of remifentanil | 90 minutes
  Occurrence of following adverse events such Drowsy, nausea, vomiting, shivering and evidence of respiratory suppression ( desaturation or bradypnea ) were documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Result] Thompson JP, Rowbotham DJ. Remifentanil--an opioid for the 21st century. Br J Anaesth. 1996 Mar;76(3):341-3. doi: 10.1093/bja/76.3.341. No abstract available. PMID 8785129
- [Result] Kaygusuz K, Yildirim A, Kol IO, Gursoy S, Mimaroglu C. Hypotensive anaesthesia with remifentanil combined with desflurane or isoflurane in tympanoplasty or endoscopic sinus surgery: a randomised, controlled trial. J Laryngol Otol. 2008 Jul;122(7):691-5. doi: 10.1017/S0022215107001545. Epub 2008 Feb 21. PMID 18289455
- [Result] Manola M, De Luca E, Moscillo L, Mastella A. Using remifentanil and sufentanil in functional endoscopic sinus surgery to improve surgical conditions. ORL J Otorhinolaryngol Relat Spec. 2005;67(2):83-6. doi: 10.1159/000084576. Epub 2005 Mar 22. PMID 15785115
- [Result] Guignard B, Bossard AE, Coste C, Sessler DI, Lebrault C, Alfonsi P, Fletcher D, Chauvin M. Acute opioid tolerance: intraoperative remifentanil increases postoperative pain and morphine requirement. Anesthesiology. 2000 Aug;93(2):409-17. doi: 10.1097/00000542-200008000-00019. PMID 10910490
- [Result] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Result] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Result] Yeom JH, Kim KH, Chon MS, Byun J, Cho SY. Remifentanil used as adjuvant in general anesthesia for spinal fusion does not exhibit acute opioid tolerance. Korean J Anesthesiol. 2012 Aug;63(2):103-7. doi: 10.4097/kjae.2012.63.2.103. Epub 2012 Aug 14. PMID 22949975
- [Result] Lee LH, Irwin MG, Lui SK. Intraoperative remifentanil infusion does not increase postoperative opioid consumption compared with 70% nitrous oxide. Anesthesiology. 2005 Feb;102(2):398-402. doi: 10.1097/00000542-200502000-00024. PMID 15681957
- [Result] Komatsu R, Turan AM, Orhan-Sungur M, McGuire J, Radke OC, Apfel CC. Remifentanil for general anaesthesia: a systematic review. Anaesthesia. 2007 Dec;62(12):1266-80. doi: 10.1111/j.1365-2044.2007.05221.x. PMID 17991265
- [Result] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Bull World Health Organ. 2007 Nov;85(11):867-72. doi: 10.2471/blt.07.045120. PMID 18038077